CLINICAL TRIAL: NCT07307131
Title: A Head-to-Head Comparison of Intralesional Furosemide-Digoxin Versus Polidocanol for the Treatment of Cutaneous Warts With 6-Month Follow-up
Brief Title: Furosemide-Digoxin vs. Polidocanol for Cutaneous Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Shams, Principal investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: intralesional treatment warts
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Warts; Human Papilloma Virus (HPV)
Keywords: Cutaneous warts, human papillomavirus, intralesional therapy, furosemide, digoxin, polidocanol, sclerotherapy
MeSH Terms: interventions — Digoxin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Furosemide and digoxin (Experimental): Intralesional combined furosemide (10 mg/ml) and digoxin (0.25 mg/ml)
  Interventions: Drug: Intralesional combined furosemide (10 mg/ml) and digoxin (0.25 mg/ml)
- Polidocanol (Active Comparator): Intralesional Polidocanol 2%
  Interventions: Drug: Intralesional polidocanol 2%

INTERVENTIONS:
Drug: Intralesional combined furosemide (10 mg/ml) and digoxin (0.25 mg/ml) — Group A (Experimental): Intralesional combined furosemide (10 mg/ml) and digoxin (0.25 mg/ml)
  Arms: Furosemide and digoxin
Drug: Intralesional polidocanol 2% — Group B (Active Comparator): Intralesional polidocanol 2%
  Arms: Polidocanol

SUMMARY:
This study compares the effectiveness and safety of two different intralesional treatments for cutaneous warts: a combination of furosemide and digoxin versus polidocanol.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, comparative clinical study to evaluate the efficacy and safety of intralesional combined furosemide-digoxin versus intralesional polidocanol in the treatment of cutaneous warts. Sixty-four adult patients were randomized to receive one of the two treatments every two weeks for a maximum of four sessions. The main goal was to see which treatment was better at completely clearing the warts. The study also looked at side effects and how often the warts came back within six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with single or multiple cutaneous warts.

Exclusion Criteria:

* History of allergies to the study medications, known cardiac or renal disease, hypertension, pregnancy or lactation, and any signs of systemic or local infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Complete Clinical Response | Up to 8 weeks
  100% clearance of the treated wart at the end of the treatment period.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Effects | Throughout the treatment period (up to 8 weeks)
  Assessment of side effects such as pain, erythema, edema, and ulceration.
Recurrence Rate | 6 months post-treatment
  Rate of wart recurrence at the 6-month follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Shams, MD, Principal Investigator — Benha University
Locations (1):
- faculty of Medicine, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No